CLINICAL TRIAL: NCT04073069
Title: Pre-emptive Scalp Infiltration With Diprospan Plus Ropivacaine for Postoperative Pain After Craniotomy in Adults
Brief Title: Scalp Infiltration With Diprospan Plus Ropivacaine for Postoperative Pain After Craniotomy in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY 2018-034-02-3
Record Dates: First submitted 2019-08-27; First posted 2019-08-28 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Pain, Postoperative; Post-Craniotomy Headache
Keywords: Postoperative Pain;; Post-Craniotomy Headache; Ropivacaine; Pre-emptive Scalp Infiltration; Diprospan
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The DR group (Experimental): Participates received peri-incisional scalp infiltration with 15ml ropivacaine 1% wt/vol, 0.5ml diprospan, plus 14.5ml saline;
  Interventions: Drug: The DR group
- The R group (Active Comparator): Participates received peri-incisional scalp infiltration with 15ml ropivacaine 1% wt/vol, plus 15ml saline;
  Interventions: Drug: The R group

INTERVENTIONS:
Drug: The DR group — Miscible liquid of diprospan and ropivacaine in this study will be peri-incisional scalp infiltration with 0.5 ml diprospan, 15 ml 1% ropivacaine and 14.5 ml normal saline miscible liquids for participants who will undergo elective craniotomy. The local infiltration solution containing will be infiltrated along the incision and throughout the entire thickness of the scalp before skin incision. The volume of local infiltration solution will be decided by surgeons according to the cut length, and the capacity of the solution will be recorded by investigator.
  Arms: The DR group
Drug: The R group — Miscible liquid of ropivacaine in this study will be peri-incisional scalp infiltration with 15 ml 1% ropivacaine and 15 ml normal saline miscible liquids for participants who will undergo elective craniotomy. The local infiltration solution containing will be infiltrated along the incision and throughout the entire thickness of the scalp before skin incision. The volume of local infiltration solution will be decided by surgeons according to the cut length, and the capacity of the solution will be recorded by investigator.
  Arms: The R group

SUMMARY:
Pain is common for the first 2 days after major craniotomy. A majority of patients would suffer from moderate-to-severe postoperative pain after undergoing craniotomy. Inadequate analgesia induced sympathetically mediated hypertension may lead to an increased risk for post-operative complications, such as arterial hypertension, intracranial hemorrhage, prolonged hospital stay, and mortality. Adequate pain control is essential for patients' prognosis and their postoperative life quality. Pain after craniotomy derives from the scalp and pericranial muscles. Local anesthetics administered around the incision have been performed clinically. However, some studies revealed that the analgesic effect of local anesthetics was not unsatisfactory due to its short pain relief duration. Pain is common for the first 2 days after major elective intracranial surgery, and the relatively short analgesic time of scalp infiltration does not seem to meet the requirements of craniotomy. Steroid such as diprospan as an adjuvant to local anesthetics intra-articular injected locally ameliorated pain intensity in knee osteoarthritis or in total knee arthroplasty. However, there has not been reported about local application of diprospan on scalp infiltration. Thus, the investigators suppose that pre-emptive scalp infiltration with steroid (diprospan) plus local anesthetic (ropivacaine) could relieve postoperative pain after craniotomy in adults.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective craniotomy for resection of tumour under general anaesthesia;
* American Society of Anesthesiologists (ASA) physical status of I , II or III;
* Participates with an anticipated fully recovery within 2 hours postoperatively.

Exclusion Criteria:

* History of craniotomy;
* Expected delayed extubation or no plan to extubate;
* Participants who cannot use a patient-controlled analgesia (PCA) device;
* Participants who cannot understand the instructions of a numeral rating scale (NRS) 35 before surgery;
* Extreme body mass index (BMI) (< 15 or > 35);
* Allergy to opioids, diprospan or ropivacaine;
* History of excessive alcohol or drug abuse, chronic opioid use (more than 2 weeks), or use of drugs with confirmed or suspected sedative or analgesic effects;
* History of psychiatric disorders, uncontrolled epilepsy or chronic headache;
* Pregnant or at breastfeeding;
* Symptomatic cardiopulmonary, renal, or liver dysfunction or history of diabetes;
* Preoperative Glasgow Coma Scale< 15;
* Suspicion of intracranial hypertension;
* Peri-incisional infection;
* Participants who have received radiation therapy and chemotherapy preoperatively or with a high probability to require a postoperative radiation therapy and chemotherapy according to the preoperative imaging.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Cumulative sufentanil consumption within 48 hours postoperatively | Within 48 hours after the operation
  All participates will receive an electronic intravenous patient-controlled analgesia (PCA) device. Participates will be advised to push the analgesic demand button if they feel pain.

SECONDARY OUTCOMES:
The number of participants who have no sufentanil consumption | Within 48 hours after the operation
  The number of participants who have not pushed the button of patient-controlled analgesia pump.
The first time to press the patient-controlled analgesia button | Within 48 hours after the operation
  The first time that the participants press the patient-controlled analgesia button.
The total times that participants press patient-controlled analgesia button | Within 48 hours postoperatively
  The total times that participants press patient-controlled analgesia button including effective presses and ineffective presses.
Numerical rating scale (NRS) | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours, 72 hours, 1 week, 2 weeks, 1 month, 3 months and 6 months after surgery
  Pain will be assessed after surgery by numerical rating scale (0 indicates no pain, 10 indicates the most severe pain imaginable).
Postoperative nausea and vomiting | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours after surgery
  Postoperative nausea and vomiting (PONV) was rated by participates as: 0, absent; 1, nausea not requiring treatment; 2, nausea requiring treatment; and 3, vomiting.
Ramsay Sedation Scale (RSS) | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours after surgery
  Ramsey 1: Anxious, agitated, restless; Ramsey 2: Cooperative, oriented, tranquil; Ramsey 3: Responsive to commands only If Asleep; Ramsey 4: Brisk response to light glabellar tap or loud auditory stimulus; Ramsey 5: Sluggish response to light glabellar tap or loud auditory stimulus; Ramsey 6: No response to light glabellar tap or loud auditory stimulus.
Respiratory depression | Within 48 hours after the operation
  Respiratory depression is defined as a respiratory rate less than 10 breaths per minute or oxygen saturation was less than ninety percent.
The times of emergency reducing blood pressure after the operation | Within 48 hours after the operation
  The criteria for treatment is determined by the participant's surgeon in charge.The times of emergency reducing blood pressure will be recording by the investigator.
Patient satisfactory scale (PSS) | t 2 hours, 4 hours, 8 hours, 24 hours, 48 hours, 72 hours, 1 week, 2 weeks, 1 month, 3 months and 6 months after surgery
  0 for unsatisfactory, and 10 for very satisfied
The total consumption of opioids during the operation | During procedure
  The total consumption of opioids during the operation
The length of stay | Approximately 2 weeks after the operation
  The duration of hospitalization after the operation
The World Health Organization Quality of Life (WHOQOL)-BREF | At 1 month, 3 months and 6 months after surgery
  Quality of life will be measured using the World Health Organisation QoL-BREF (WHOQOL-BREF) questionnaire. The WHOQOL-BREF is a abbreviated version of the WHOQOL-100 assessment. WHOQOL-BREF is a self-report questionnaire that contains 26 items and addresses 4 QOL domains: physical health (7 items), psychological health (6 items), social relationships (3 items) and environment (8 items). Two other items measure overall QOL and general health. Each domain's mean score can range between 4 and 20 and a higher score indicates a higher quality of life. The mean score of items within each domain is used to calculate the domain score. A transformation method converts domain scores to a 0-100 scale.
Wound Healing Score | At 1 month after surgery
  Skin Healing 1: fully healed; 2: ≤3 cm in total not healed; 3: >3 cm not healed; 4: areas of necrosis ≤3 cm; 5: areas of necrosis >3 cm Infection 1: none; 2: ≤0.5-cm margin of redness; 3: more redness or superficial pus; 4: deep infection; not applicable Hair Regrowth 1: even regrowth along wound; 2: ≤3 cm not regrowing; 3: >3-6 cm not regrowing; 4: >6 cm not regrowing; not applicable

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gottschalk A, Berkow LC, Stevens RD, Mirski M, Thompson RE, White ED, Weingart JD, Long DM, Yaster M. Prospective evaluation of pain and analgesic use following major elective intracranial surgery. J Neurosurg. 2007 Feb;106(2):210-6. doi: 10.3171/jns.2007.106.2.210. PMID 17410701
- [Background] Dunn LK, Naik BI, Nemergut EC, Durieux ME. Post-Craniotomy Pain Management: Beyond Opioids. Curr Neurol Neurosci Rep. 2016 Oct;16(10):93. doi: 10.1007/s11910-016-0693-y. PMID 27604271
- [Background] Chaki T, Sugino S, Janicki PK, Ishioka Y, Hatakeyama Y, Hayase T, Kaneuchi-Yamashita M, Kohri N, Yamakage M. Efficacy and Safety of a Lidocaine and Ropivacaine Mixture for Scalp Nerve Block and Local Infiltration Anesthesia in Patients Undergoing Awake Craniotomy. J Neurosurg Anesthesiol. 2016 Jan;28(1):1-5. doi: 10.1097/ANA.0000000000000149. PMID 25493926
- [Background] Romsing J, Moiniche S, Ostergaard D, Dahl JB. Local infiltration with NSAIDs for postoperative analgesia: evidence for a peripheral analgesic action. Acta Anaesthesiol Scand. 2000 Jul;44(6):672-83. doi: 10.1034/j.1399-6576.2000.440607.x. PMID 10903014
- [Background] Nakai T, Tamaki M, Nakamura T, Nakai T, Onishi A, Hashimoto K. Controlling pain after total knee arthroplasty using a multimodal protocol with local periarticular injections. J Orthop. 2013 Mar 17;10(2):92-4. doi: 10.1016/j.jor.2013.02.001. eCollection 2013. PMID 24403757
- [Background] Watanabe K, Tokumine J, Yorozu T, Moriyama K, Sakamoto H, Inoue T. Particulate-steroid betamethasone added to ropivacaine in interscalene brachial plexus block for arthroscopic rotator cuff repair improves postoperative analgesia. BMC Anesthesiol. 2016 Oct 4;16(1):84. doi: 10.1186/s12871-016-0251-9. PMID 27716229